CLINICAL TRIAL: NCT06462014
Title: Description of Relugolix Use in Patients With Prostate Cancer: An Analysis of National Veterans Affairs Health Care Network Data
Brief Title: Description of Relugolix Use in Patients With Prostate Cancer Within the VHA
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4751009; VHA Study (Other: Alias Study Number)
Record Dates: First submitted 2024-05-23; First posted 2024-06-17 (Actual); Results first posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
Keywords: Relugolix
MeSH Terms: conditions — Prostatic Neoplasms | interventions — relugolix

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Relugolix patients: Patients who have initiated relugolix
  Interventions: Drug: Relugolix

INTERVENTIONS:
Drug: Relugolix — relugolix

SUMMARY:
The purpose of this real-world study is the learn about the demographics and clinical characteristics of patients with prostate cancer who initiated relugolix

DETAILED DESCRIPTION:
Prostate cancer (PC) is the most common cancer and the second leading cause of cancer death among men in the United States. Androgen deprivation therapy (ADT) such as injectable luteinizing hormone-releasing hormone (LHRH) agonists (e.g., leuprolide) is the standard of care for PC patients. ADT treatment can suppress testosterone level to castrate level and delay the progression of the disease.

Relugolix is a recently approved oral GnRH antagonist. While the introduction of relugolix has offered a unique opportunity for patients with PC, it's vital to understand how it is being used in real-world.

ELIGIBILITY:
Inclusion Criteria:

* Male with ≥ 1 diagnosis for PC
* Had ≥ 2 prescriptions of relugolix on or after the first observed PC diagnosis.
* Index date: the initiation date of relugolix
* At least 18 years old at the index date

Exclusion Criteria:

* had surgical castration (bilateral orchiectomy) any time before the index date

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients with prostate cancer
Study Population: Men who are part of this study initiated relugolix as part of their usual treatment for PC
Sampling Method: Non-Probability Sample
Enrollment: 507 (Actual)
Dates: Start 2024-06-19 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Freedland SJ, Ramaswamy K, Kavati A, Gao W, Razo JF, Cole M, Li B, Yang H, Guo T, Chen G, McKay RR. Retrospective Analysis of Racial Differences in Treatment Patterns and Prostate-Specific Antigen Responses Among Patients with Prostate Cancer Treated with Relugolix in the Veterans Health Administration. Adv Ther. 2025 Dec;42(12):6278-6294. doi: 10.1007/s12325-025-03390-6. Epub 2025 Nov 1. PMID 41174189
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4751009

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data from participants with a diagnosis of prostate cancer between 01-Jan-2006 to 31-Dec-2023 and who had initiated relugolix anytime between 18-Dec-2020 (approval date for relugolix in the United States) to 31-Dec-2023 was included. Data was collected from the National Veterans Affairs (VA) Health Care Network database. Available retrospective data was evaluated over 178 days (from 19-Jun-2024 to 13-Dec-2024) in this observational study per its objective.
Groups:
- Relugolix: Participants who were diagnosed with prostate cancer and had initiated relugolix between 18-Dec-2020 to 31-Dec-2023 were observed. No intervention was administered in this study.
Period: Overall Study
Arm/Group | Relugolix
Started | 507
Completed | 507
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Relugolix
Number analyzed (Participants) | 507
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.2 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 507
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 313
  Black | 141
  Hispanic | 16
  Other | 6
  Unknown | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants According to Geographic Region
Description: The number of participants according to geographic regions of the United States (South, West, Northeast and Midwest) as documented during baseline period were reported in this outcome measure. Baseline period was 1 year prior to index date; index date was the initiation date of relugolix (anytime between 18-Dec-2020 to 31-Dec-2023) on or after the first observed prostate cancer diagnosis.
Time Frame: Baseline period = Up to 1 year prior to index date; available data observed retrospectively over 178 days in this study
Population: Analysis population included all eligible participants whose data was retrieved and observed in this retrospective observational study.
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix
Number analyzed (Participants) | 507
Participants
  South | 240
  West | 94
  Northeast | 93
  Midwest | 80

2. Primary Outcome: Number of Participants According to Index Year
Description: Number of participants according to index year (2020, 2021, 2022 and 2023) were reported in this outcome measure. The index date was defined as the initiation date of relugolix (anytime between 18-Dec-2020 to 31-Dec-2023) on or after the first observed prostate cancer diagnosis.
Time Frame: At Index date (anytime between 18-Dec-2020 to 31-Dec- 2023 [approximately 3 years]; available data observed retrospectively over 178 days in this study
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix
Number analyzed (Participants) | 507
Participants
  2020 | 0
  2021 | 81
  2022 | 203
  2023 | 223

3. Primary Outcome: Time From First Observed Prostate Cancer Diagnosis Date to the Index Date
Description: Time from the first observed prostate cancer date to the index date was evaluated. All data available prior to the index date were used. The index date was defined as the initiation date of relugolix (anytime between 18-Dec-2020 to 31-Dec-2023) on or after the first observed prostate cancer diagnosis. Participants with a diagnosis of prostate cancer between 01-Jan-2006 to 31-Dec-2023 were considered.
Time Frame: From prostate cancer diagnosis to index date (approximately maximum up to 18 years); available data observed retrospectively over 178 days in this study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Relugolix
Number analyzed (Participants) | 507
Months | 55.8 (61.7)

4. Primary Outcome: Number of Participants According to Type of Previous Treatments Received
Description: Number of participants according to treatments received previously such as pain medication, androgen receptor pathway inhibitor, androgen deprivation therapy, chronic oral corticosteroid use, non-steroidal anti-androgen, radiotherapy, olaparib, prostatectomy and chemotherapy in the baseline period were reported in this outcome measure. Baseline period was 1 year prior to index date; index date was the initiation date of relugolix (anytime between 18-Dec-2020 to 31-Dec-2023) on or after the first observed prostate cancer diagnosis. One participant could have received more than 1 treatment.
Time Frame: Baseline period = Up to 1 year prior to index date; available data observed retrospectively over 178 days in this study
Population: Analysis population included all eligible participants whose data was retrieved and observed in this retrospective observational study. All the participants of the study were analyzed but not all participants might have contributed to the data reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix
Number analyzed (Participants) | 507
Participants
  Pain medication | 103
  Androgen receptor pathway inhibitor | 86
  Androgen deprivation therapy | 77
  Chronic oral corticosteroid use | 48
  Non-steroidal anti-androgen | 46
  Radiotherapy | 7
  Olaparib | 3
  Prostatectomy | 3
  Chemotherapy | 2

5. Primary Outcome: Number of Participants According to Metastasis Status
Description: Number of participants according to metastasis status (metastatic prostate cancer and non-metastatic prostate cancer) were reported in this outcome measure. Metastatic prostate cancer was defined as having evidence of during the baseline period or within 90 days after the index date. Baseline period was 1 year prior to index date; index date was the initiation date of relugolix (anytime between 18-Dec-2020 to 31-Dec-2023) on or after the first observed prostate cancer diagnosis.
Time Frame: Baseline period = Up to 1 year prior to index date or within 90 days after the index date; available data observed retrospectively over 178 days in this study
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix
Number analyzed (Participants) | 507
Participants
  Metastatic prostate cancer | 169
  Non-metastatic prostate cancer | 338

6. Primary Outcome: Number of Participants According to Site of Metastasis
Description: Number of participants with a metastatic diagnosis at the sites: bone only, node only, bone and node, viscera and other (urinary organs, genital organs, skin, kidney, adrenal, brain, spinal, and other nervous system), were reported among participants with metastatic prostate cancer. Metastatic prostate cancer was defined as having evidence of metastasis any time prior to the index date or within 90 days after the index date. Baseline period was 1 year prior to index date; index date was the initiation date of relugolix (anytime between 18-Dec-2020 to 31-Dec-2023) on or after the first observed prostate cancer diagnosis.
Time Frame: as for outcome 5
Population: Analysis population included all eligible participants whose data was retrieved and observed in this retrospective observational study. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix
Number analyzed (Participants) | 169
Participants
  Bone only | 59
  Node only | 34
  Bone and Node | 20
  Viscera | 20
  Other | 36

7. Primary Outcome: Number of Participants According to Androgen Deprivation Therapy (ADT) Status
Description: ADT naïve was defined as having no records of any systemic ADT ever based on all available data prior to the index date (i.e., including baseline period data and any available data prior to the baseline period). Systemic ADT included luteinizing hormone-releasing hormone (LHRH) agonists and gonadotropin-releasing hormone (GnRH) antagonists (i.e., degarelix, relugolix, goserelin, histrelin, leuprolide, triptorelin). ADT experienced was defined as having any records of systemic ADT based on all available data prior to the index date (i.e., including baseline period data and any available data prior to the baseline period). Baseline period was 1 year prior to index date; index date was the initiation date of relugolix (anytime between 18-Dec-2020 to 31-Dec-2023) on or after the first observed prostate cancer diagnosis.
Time Frame: Any time prior to index date including baseline period (approximately maximum up to 18 years); available data observed retrospectively over 178 days in this study
Population: Analysis population included all eligible participants whose data was retrieved and observed in this retrospective observational study. Here, "Number Analyzed" signifies number of participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix
Number analyzed (Participants) | 507
Participants
  Metastatic PC: number analyzed (Participants) | 169
  Metastatic PC: ADT naïve | 80
  Metastatic PC: ADT experienced | 89
  No known metastases: number analyzed (Participants) | 338
  No known metastases: ADT naïve | 286
  No known metastases: ADT experienced | 52

8. Primary Outcome: Prostate-Specific Antigen (PSA) Value at 180 Days Prior to Index Date
Description: The index date was defined as the initiation date of relugolix (anytime between 18-Dec-2020 to 31-Dec-2023) on or after the first observed PC diagnosis.
Time Frame: 180 days prior to Index date; data observed retrospectively over 178 days in this study
Population: Analysis population included all eligible participants whose data was retrieved and observed in this retrospective observational study. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Relugolix
Number analyzed (Participants) | 313
Nanograms per milliliter | 118.8 (1080.6)

9. Primary Outcome: Testosterone Value at 180 Days Prior to Index Date
Description: as for outcome 8
Time Frame: 180 days prior to Index date; data observed retrospectively over 178 days in this study
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Nanograms per deciliter
Arm/Group | Relugolix
Number analyzed (Participants) | 109
Nanograms per deciliter | 200.9 (213.1)

10. Primary Outcome: Mean National Cancer Institute (NCI) Charlson Comorbidity Index (CCI) Score
Description: CCI based on various comorbid conditions such as myocardial infarction, congestive heart failure, peripheral vascular disease, cerebrovascular disease, dementia, chronic obstructive pulmonary disease, rheumatologic disease, peptic ulcer disease, mild liver disease, diabetes (mild to moderate), diabetes + complications, hemiplegia or paraplegia, renal disease, any malignancy (lymphoma and leukemia), moderate/severe liver disease, metastatic solid tumor, and acquired immune deficiency syndrome (AIDS) were reported. CCI score range was from 0 to 14, where "0"= low comorbid condition and "14"= high comorbid condition, higher scores indicated more comorbidity. Baseline period was 1 year prior to index date; index date was the initiation date of relugolix (anytime between 18-Dec-2020 to 31-Dec-2023) on or after the first observed prostate cancer diagnosis.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Relugolix
Number analyzed (Participants) | 507
Units on a scale | 1.8 (2.1)

11. Primary Outcome: Number of Participants According to Comorbidities
Description: Number of participants according to comorbidities (hypertension, hyperlipidemia, diabetes, major adverse cardiovascular event, depression, congestive heart failure, sexual dysfunction, chronic obstructive pulmonary disease, anxiety, cognitive impairment, urinary tract infection, myocardial infarction, arrhythmia, stroke, acute coronary syndrome, angina pectoris, inflammatory bowel disease, hot flashes) were reported in this outcome measure. Baseline period was 1 year prior to index date; index date was the initiation date of relugolix (anytime between 18-Dec-2020 to 31-Dec-2023) on or after the first observed prostate cancer diagnosis. One participant could have more than one comorbidity.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix
Number analyzed (Participants) | 507
Participants
  Hypertension | 357
  Hyperlipidemia | 319
  Diabetes | 168
  Major adverse cardiovascular event | 114
  Depression | 90
  Congestive heart failure | 74
  Sexual dysfunction | 74
  Chronic obstructive pulmonary disease | 68
  Anxiety | 57
  Cognitive impairment | 57
  Urinary tract infection | 52
  Myocardial infarction | 31
  Arrhythmia | 28
  Stroke | 26
  Acute coronary syndrome | 15
  Angina pectoris | 11
  Inflammatory bowel disease | 6
  Hot flashes | 2

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed on and after index-date till the end of continuous eligibility, data availability, or death, whichever occurred first (maximum follow-up on and after index date was of 19.7 months). Time frame was not applicable for adverse events as adverse events were not planned to be monitored and evaluated for the study.
Description: Due to non-interventional nature of the study and nature of data sources, the minimum criteria for reporting an adverse event (i.e., identifiable participant, identifiable reporter, a suspect product, and event) could not be met, hence adverse events were not planned to be monitored and evaluated (thus at risk appears "0").
Arm/Group | Relugolix
All-Cause Mortality (participants affected / at risk) | 38/507
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-15): https://cdn.clinicaltrials.gov/large-docs/14/NCT06462014/Prot_SAP_000.pdf